CLINICAL TRIAL: NCT01263925
Title: Intravenous Prostaglandin E1 Treatment in Outpatients With Intermittent Claudication
Brief Title: Prostaglandin E1 in Outpatients With Intermittent Claudication
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SP0580
Record Dates: First submitted 2010-12-17; First posted 2010-12-21 (Estimated); Results first posted 2012-06-29 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2012-05

CONDITIONS: Stage II Peripheral Arterial Occlusive Disease; Intermittent Claudication Fontaine Stage II PAOD
Keywords: Alprostadil; Prostaglandin E1; Prostavasin®; PAOD
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1 | interventions — Alprostadil; Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alprostadil (Experimental): Alprostadil (Prostaglandin E1) intravenous and matching Placebo to Pentoxifylline oral
  Interventions: Drug: Alprostadil (Prostaglandin E1); Drug: Placebo to Pentoxifylline oral
- Pentoxifylline (Active Comparator): Pentoxifylline oral and matching Placebo to Alprostadil (Prostaglandin E1) intravenous
  Interventions: Drug: Pentoxifylline; Drug: Placebo to Alprostadil (Prostaglandin E1) intravenous

INTERVENTIONS:
Drug: Alprostadil (Prostaglandin E1) — 4-week Daily Treatment Period 1: 4 weeks of 1 x daily intravenous infusion of 3 ampoules (20 µg) of Prostaglandin E1 (total 60 µg) in 50 - 250 ml physiological saline solution over 2 hours.
  4-week Interval Treatment Period 2: 4 weeks of 2 x weekly intravenous infusion of 3 ampoules (20 µg) of Prostaglandin E1 (total 60 µg) in 50 - 250 ml physiological saline solution over 2 hours.
  Other Names: Prostavasin
  Arms: Alprostadil
Drug: Pentoxifylline — 4-week Daily Treatment Period 1: 4 weeks of 2 x daily (including weekends) 600 mg Pentoxifylline tablets.
  4-week Interval Treatment Period 2: 4 weeks of 2 x daily (including weekends) 600 mg Pentoxifylline tablets.
  Other Names: Trental®
  Arms: Pentoxifylline
Drug: Placebo to Pentoxifylline oral — 4-week Daily Treatment Period 1: 4 weeks of 2 x daily (including weekends) matching Placebo to Pentoxifylline tablets.
  4-week Interval Treatment Period 2: 4 weeks of 2 x daily (including weekends) matching Placebo to Pentoxifylline tablets.
  Arms: Alprostadil
Drug: Placebo to Alprostadil (Prostaglandin E1) intravenous — 4-week Daily Treatment Period 1: 4 weeks of 1 x daily intravenous infusion of Placebo in 50 - 250 ml physiological saline solution over 2 hours.
  4-week Interval Treatment Period 2: 4 weeks of 2 x weekly intravenous infusion of Placebo in 50 - 250 ml physiological saline solution over 2 hours.
  Arms: Pentoxifylline

SUMMARY:
Investigate, under outpatient conditions, both the effect of 4 weeks of daily treatment with Prostaglandin E1 and that of 4 weeks of interval treatment (two infusions per week) on the pain-free walking distance in patients with Intermittent Claudication.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Peripheral Arterial Occlusive Disease (PAOD) of the lower extremity in Fontaine stage II
* Maximum walking distance on the treadmill (12 %, 3 km/h) between 30 and 150 m
* Stable Intermittent Claudication of at least 6 months standing with no acute shortening of walking distance over the past 3 months
* Stenoses or occlusions below the Femoral Bifurcation (above-knee or below-knee type) confirmed by duplex US or angiography
* Ankle/brachial index ≤ 0.90 with a decrease in systolic ankle pressure of ≥ 10 % after maximum loading (maximum walking distance on the treadmill at 3 km/h, 12 %)
* The patient is physically and mentally capable of participating in the trial
* Patient age > 40 years, male and female
* Patient is informed and given ample time and opportunity to think about her/his participation and has given her/his written informed consent
* Patient is willing and able to comply with all trial requirements

Exclusion Criteria:

* Surgical or other interventional measures performed on the affected extremity and Prostaglandin treatment within the 6 months immediately prior to the trial
* Rest pain and Necroses
* Systolic ankle pressure less than 50 mmHg
* Change in maximum walking distance during the one-week Run-in Phase of more than ± 25 % of Baseline
* Successful physical walking training within the 6 months immediately prior to the trial
* Inflammatory vascular diseases
* Polyneuropathy in Diabetes Mellitus
* Diseases limiting walking distance (Arthrosis, inflammatory diseases of the joints, neurological disease, diseases of the Vertebral Column, cardiopulmonary diseases)
* History of Pulmonary Oedema
* Myocardial infarction within the past 6 months
* Pregnancy or nursing
* Known hypersensitivity to any components of the trial medication or comparative drug
* Renal insufficiency, compensated retention (creatinine > 2.0 mg/dL)
* Severe retinal Haemorrhage
* Massive Haemorrhage
* Known existing malignant diseases
* Vasoactive concomitant medication (e.g. Naftidrofuryl, Pentoxifylline, Buflomedil, Cilostazol), or other Prostaglandins
* Untreated or uncontrolled Hypertension (systolic blood pressure ≥ 180 mmHg, diastolic blood pressure ≥ 110 mmHg)
* Previous participation of the patient in the present trial
* Participation of the patient in a trial with the same objectives within the past 6 months, or is currently participating in another trial
* Illness of the patient due to alcohol or drug-abuse within the past 6 months
* Serious illness of the patient that the investigator considers to compromise his/her participation in the trial

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 561 (Actual)
Dates: Start 2001-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (36):
- Germany (36):
  - Aachen
  - Bad Säckingen
  - Berlin
  - Bottrop
  - Cologne
  - Dortmund
  - Dresden
  - Düsseldorf
  - Essen
  - Essen-Steele
  - Freiburg im Breisgau
  - Gaggenau
  - Görlitz
  - Hamburg
  - Hanover
  - Hattingen
  - Heidelberg
  - Homburg
  - Jena
  - Karlsbad-Lang Ensteinbach
  - Kassel
  - Krefeld
  - Leipzig
  - Lüneburg
  - Mannheim
  - Mannheim-Lindenhof
  - Mönchengladbach
  - München
  - Neuss
  - Nuremberg
  - Osnabrück
  - Papenburg
  - Regensburg
  - Seesen
  - Warendorf
  - Wuppertal

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 607 screened subjects, 561 have been randomized. Of these 561 randomized subjects, 541 are included in the Full Analysis Set (FAS). FAS includes all randomized subjects who received at least one dose of trial medication and who have at least one valid measurement of pain-free walking distance under therapy.
Pre-assignment Details: Participant Flow shows all randomized subjects. Baseline Characteristics refer to the FAS.
Groups:
- Alprostadil: 4-week Daily Treatment Period 1: 4 weeks of 1 x daily intravenous infusion of 3 ampoules (20 μg) of Prostaglandin E1 (total 60 μg) in 50 - 250 ml physiological saline solution over 2 hours and in addition 2 x daily (including weekends) Placebo tablets.
  4-week Interval Treatment Period 2: 4 weeks of 2 x weekly intravenous infusion of 3 ampoules (20 μg) of Prostaglandin E1 (total 60 μg) in 50 - 250 ml physiological saline solution over 2 hours and in addition 2 x daily (including weekends) Placebo tablets.
- Pentoxifylline: 4-week Daily Treatment Period 1: 4 weeks of 1 x daily intravenous infusion of Placebo in 50 - 250 ml physiological saline solution over 2 hours and in addition 2 x daily (including weekends) 600 mg Pentoxifylline tablets.
  4-week Interval Treatment Period 2: 4 weeks of 2 x weekly intravenous infusion of Placebo in 50 - 250 ml physiological saline solution over 2 hours and in addition 2 x daily (including weekends) 600 mg Pentoxifylline tablets.
Period: Overall Study
Arm/Group | Alprostadil | Pentoxifylline
Started | 276 | 285
Full Analysis Set | 269 | 272
Completed | 225 | 233
Not Completed | 51 | 52
Not completed — Protocol Violation | 1 | 0
Not completed — Lack of Efficacy | 0 | 1
Not completed — Adverse Event | 23 | 22
Not completed — Unsatisfactory Compliance of Subject | 8 | 5
Not completed — Withdrawal by Subject | 6 | 8
Not completed — Other | 4 | 4
Not completed — Lost to Follow-up | 3 | 1
Not completed — Lack of Efficacy/ Adverse Event (AE) | 1 | 1
Not completed — AE/ Unsatisfactory Compliance | 2 | 2
Not completed — AE/ Withdrawal | 1 | 4
Not completed — Unsatisfactory Compliance/ Withdrawal | 1 | 1
Not completed — Unsatisfactory Compl./ Lost to Follow up | 1 | 2
Not completed — Withdrawal/ Not specified | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alprostadil | Pentoxifylline | Total
Number analyzed (Participants) | 269 | 272 | 541
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (8.6) | 66.8 (8.8) | 66.5 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 89 | 173
  Male | 185 | 183 | 368
Ethnicity [Number; unit: participants]
  Caucasian | 269 | 271 | 540
  Asian | 0 | 1 | 1
Age categories [Number; unit: participants]
  >18 - <65 | 108 | 100 | 208
  >=65 - <75 | 114 | 119 | 233
  >=75 | 47 | 53 | 100
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 77.8 (13.9) | 77.9 (13.5) | 77.9 (13.7)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 170.2 (8.6) | 169.3 (8.6) | 169.7 (8.6)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram/ meter^2 (kg/m^2)] | 26.77 (3.87) | 27.11 (3.75) | 26.94 (3.81)
Duration of Primary Disease [Mean (Standard Deviation); unit: years] | 4.9 (5.1) | 4.3 (4.4) | 4.6 (4.8)

OUTCOME MEASURES:

1. Primary Outcome: Ratio of Pain-free Walking Distance After Period 2 in Comparison With the Findings at Baseline
Description: The ratio of pain-free walking distance was calculated by the pain-free walking distance after Period 2 divided by the pain-free walking distance at Baseline with determination of pain-free walking distances on the treadmill (12 % grade and 3 km/h). If a subject was not familiar with the treadmill, at least two test determinations were performed to accustom him/her to the treadmill. For all treadmill determinations the subject has been prevented from observing the treadmill display of the walking distance achieved.
Time Frame: From Baseline to the end of 4 weeks of Interval Treatment (Period 2)
Population: Full Analysis Set (FAS).
Measure: Mean (Standard Deviation); unit: meter/meter
Arm/Group | Alprostadil | Pentoxifylline
Number analyzed (Participants) | 269 | 272
meter/meter | 2.60 (12.22) [1.1 to 4.1] | 1.98 (3.61)

2. Primary Outcome: Ratio of Pain-free Walking Distance After Period 3 in Comparison With the Findings at Baseline
Description: The ratio of pain-free walking distance was calculated by the pain-free walking distance after Period 3 divided by the pain-free walking distance at Baseline with determination of pain-free walking distances on the treadmill (12 % grade and 3 km/h). If a subject was not familiar with the treadmill, at least two test determinations were performed to accustom him/her to the treadmill. For all treadmill determinations the subject has been prevented from observing the treadmill display of the walking distance achieved.
Time Frame: From Baseline to the end of 6-months Follow-up (Period 3)
Population: Full Analysis Set (FAS).
Measure: Mean (Standard Deviation); unit: meter/meter
Arm/Group | Alprostadil | Pentoxifylline
Number analyzed (Participants) | 269 | 272
meter/meter | 2.27 (3.00) | 2.36 (2.69)

3. Primary Outcome: Ratio of Pain-free Walking Distance After Period 1 in Comparison With the Findings at Baseline
Description: The ratio of pain-free walking distance was calculated by the pain-free walking distance after Period 1 divided by the pain-free walking distance at Baseline with determination of pain-free walking distances on the treadmill (12 % grade and 3 km/h). If a subject was not familiar with the treadmill, at least two test determinations were performed to accustom him/her to the treadmill. For all treadmill determinations the subject has been prevented from observing the treadmill display of the walking distance achieved.
Time Frame: From Baseline to the end of 4 weeks of Daily Treatment (Period 1)
Population: Full Analysis Set (FAS).
Measure: Mean (Standard Deviation); unit: meter/meter
Arm/Group | Alprostadil | Pentoxifylline
Number analyzed (Participants) | 269 | 272
meter/meter | 1.58 (1.92) | 1.58 (2.59)

4. Secondary Outcome: Ratio of Pain-free Walking Distance After Period 2 in Comparison With the Findings After Period 1
Description: The ratio of pain-free walking distance was calculated by the pain-free walking distance after Period 2 divided by the pain-free walking distance after Period 1 with determination of pain-free walking distances on the treadmill (12 % grade and 3 km/h). If a subject was not familiar with the treadmill, at least two test determinations were performed to accustom him/her to the treadmill. For all treadmill determinations the subject has been prevented from observing the treadmill display of the walking distance achieved.
Time Frame: From the end of 4 weeks of Daily Treatment (Period 1) to the end of 4 weeks of Interval Treatment (Period 2)
Population: Full Analysis Set (FAS).
Measure: Mean (Standard Deviation); unit: meter/meter
Arm/Group | Alprostadil | Pentoxifylline
Number analyzed (Participants) | 269 | 272
meter/meter | 1.25 (0.64) | 1.24 (0.50)

5. Secondary Outcome: Ratio of Pain-free Walking Distance After Period 3 in Comparison With the Findings After Period 1
Description: The ratio of pain-free walking distance was calculated by the pain-free walking distance after Period 3 divided by the pain-free walking distance after Period 1 with determination of pain-free walking distances on the treadmill (12 % grade and 3 km/h). If a subject was not familiar with the treadmill, at least two test determinations were performed to accustom him/her to the treadmill. For all treadmill determinations the subject has been prevented from observing the treadmill display of the walking distance achieved.
Time Frame: From the end of 4 weeks of Daily Treatment (Period 1) to the end of 6-months Follow-up (Period 3)
Population: Full Analysis Set (FAS).
Measure: Mean (Standard Deviation); unit: meter/meter
Arm/Group | Alprostadil | Pentoxifylline
Number analyzed (Participants) | 269 | 272
meter/meter | 1.54 (1.53) | 1.57 (1.10)

6. Secondary Outcome: Ratio of Pain-free Walking Distance After Period 3 in Comparison With the Findings After Period 2
Description: The ratio of pain-free walking distance was calculated by the pain-free walking distance after Period 3 divided by the pain-free walking distance after Period 2 with determination of pain-free walking distances on the treadmill (12 % grade and 3 km/h). If a subject was not familiar with the treadmill, at least two test determinations were performed to accustom him/her to the treadmill. For all treadmill determinations the subject has been prevented from observing the treadmill display of the walking distance achieved.
Time Frame: From the end of 4 weeks of Interval Treatment (Period 2) to the end of 6-months Follow-up (Period 3)
Population: Full Analysis Set (FAS).
Measure: Mean (Standard Deviation); unit: meter/meter
Arm/Group | Alprostadil | Pentoxifylline
Number analyzed (Participants) | 269 | 272
meter/meter | 1.26 (0.85) | 1.28 (0.74)

7. Secondary Outcome: Ratio of Maximum Walking Distance After Period 1 in Comparison With the Findings at Baseline
Description: The ratio of maximum walking distance was calculated by the maximum walking distance after Period 1 divided by the maximum walking distance at Baseline with determination of maximum walking distances on the treadmill (12 % grade and 3 km/h). If a subject was not familiar with the treadmill, at least two test determinations were performed to accustom him/her to the treadmill. For all treadmill determinations the subject has been prevented from observing the treadmill display of the walking distance achieved.
Time Frame: From Baseline to the end of 4 weeks of Daily Treatment (Period 1)
Population: Full Analysis Set (FAS).
Measure: Mean (Standard Deviation); unit: meter/meter
Arm/Group | Alprostadil | Pentoxifylline
Number analyzed (Participants) | 269 | 272
meter/meter | 1.39 (0.53) | 1.43 (1.34)

8. Secondary Outcome: Ratio of Maximum Walking Distance After Period 2 in Comparison With the Findings at Baseline
Description: The ratio of maximum walking distance was calculated by the maximum walking distance after Period 2 divided by the maximum walking distance at Baseline with determination of maximum walking distances on the treadmill (12 % grade and 3 km/h). If a subject was not familiar with the treadmill, at least two test determinations were performed to accustom him/her to the treadmill. For all treadmill determinations the subject has been prevented from observing the treadmill display of the walking distance achieved.
Time Frame: From Baseline to the end of 4 weeks of Interval Treatment (Period 2)
Population: Full Analysis Set (FAS).
Measure: Mean (Standard Deviation); unit: meter/meter
Arm/Group | Alprostadil | Pentoxifylline
Number analyzed (Participants) | 269 | 272
meter/meter | 1.64 (0.86) | 1.76 (1.78)

9. Secondary Outcome: Ratio of Maximum Walking Distance After Period 2 in Comparison With the Findings After Period 1
Description: The ratio of maximum walking distance was calculated by the maximum walking distance after Period 2 divided by the maximum walking distance after Period 1 with determination of maximum walking distances on the treadmill (12 % grade and 3 km/h). If a subject was not familiar with the treadmill, at least two test determinations were performed to accustom him/her to the treadmill. For all treadmill determinations the subject has been prevented from observing the treadmill display of the walking distance achieved.
Time Frame: From the end of 4 weeks of Daily Treatment (Period 1) to the end of 4 weeks of Interval Treatment (Period 2)
Population: Full Analysis Set (FAS).
Measure: Mean (Standard Deviation); unit: meter/meter
Arm/Group | Alprostadil | Pentoxifylline
Number analyzed (Participants) | 269 | 272
meter/meter | 1.20 (0.50) | 1.21 (0.41)

10. Secondary Outcome: Ratio of Maximum Walking Distance After Period 3 in Comparison With the Findings at Baseline
Description: The ratio of maximum walking distance was calculated by the maximum walking distance after Period 3 divided by the maximum walking distance at Baseline with determination of maximum walking distances on the treadmill (12 % grade and 3 km/h). If a subject was not familiar with the treadmill, at least two test determinations were performed to accustom him/her to the treadmill. For all treadmill determinations the subject has been prevented from observing the treadmill display of the walking distance achieved.
Time Frame: From Baseline to the end of 6-months Follow-up (Period 3)
Population: Full Analysis Set (FAS).
Measure: Mean (Standard Deviation); unit: meter/meter
Arm/Group | Alprostadil | Pentoxifylline
Number analyzed (Participants) | 269 | 272
meter/meter | 1.89 (1.40) | 1.99 (1.61)

11. Secondary Outcome: Ratio of Maximum Walking Distance After Period 3 in Comparison With the Findings After Period 1
Description: The ratio of maximum walking distance was calculated by the maximum walking distance after Period 3 divided by the maximum walking distance after Period 1 with determination of maximum walking distances on the treadmill (12 % grade and 3 km/h). If a subject was not familiar with the treadmill, at least two test determinations were performed to accustom him/her to the treadmill. For all treadmill determinations the subject has been prevented from observing the treadmill display of the walking distance achieved.
Time Frame: From the end of 4 weeks of Daily Treatment (Period 1) to the end of 6-months Follow-up (Period 3)
Population: Full Analysis Set (FAS).
Measure: Mean (Standard Deviation); unit: meter/meter
Arm/Group | Alprostadil | Pentoxifylline
Number analyzed (Participants) | 269 | 272
meter/meter | 1.39 (0.87) | 1.42 (0.80)

12. Secondary Outcome: Ratio of Maximum Walking Distance After Period 3 in Comparison With the Findings After Period 2
Description: The ratio of maximum walking distance was calculated by the maximum walking distance after Period 3 divided by the maximum walking distance after Period 2 with determination of maximum walking distances on the treadmill (12 % grade and 3 km/h). If a subject was not familiar with the treadmill, at least two test determinations were performed to accustom him/her to the treadmill. For all treadmill determinations the subject has been prevented from observing the treadmill display of the walking distance achieved.
Time Frame: From the end of 4 weeks of Interval Treatment (Period 2) to the end of 6-months Follow-up (Period 3)
Population: Full Analysis Set (FAS).
Measure: Mean (Standard Deviation); unit: meter/meter
Arm/Group | Alprostadil | Pentoxifylline
Number analyzed (Participants) | 269 | 272
meter/meter | 1.18 (0.58) | 1.17 (0.50)

13. Secondary Outcome: Changes in Quality of Life (as Measured With the PAVK 86 Questionnaire) From Baseline to the End of Period 1
Description: Scores for subscales were calculated by summing non-missing item scores ranging from 1 (not at all; best possible outcome) to 4 (extremely; worst possible outcome) divided by the number of non-missing items. Hence each subscale score ranges from 1 (best possible outcome) to 4 (worst possible outcome). For subscales 'Mood' and 'Treatment expectation' five items each had to be reversed in order. Additionally, subjects were asked to assess their general health and quality of life on an ordinal scale between 0 (very good) and 10 (very poor).
  Negative changes show a decrease from Baseline.
Time Frame: From Baseline to the end of 4 weeks of Daily Treatment (Period 1)
Population: Full Analysis Set (FAS). For each subscale of the questionnaire, Mean and SD are presented for non-missing values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alprostadil | Pentoxifylline
Number analyzed (Participants) | 269 | 272
units on a scale
  Pain | -0.24 (0.44) | -0.27 (0.49)
  Functional status | -0.21 (0.40) | -0.18 (0.41)
  Anxiety | -0.16 (0.51) | -0.18 (0.54)
  Mood | -0.07 (0.34) | -0.08 (0.37)
  Social life | -0.05 (0.34) | -0.02 (0.33)
  Expectation of treatment | -0.00 (0.42) | 0.01 (0.42)
  State of general health during the last week | -0.51 (1.48) | -0.36 (1.60)
  Quality of life during the last week | -0.37 (1.58) | -0.38 (1.78)

14. Secondary Outcome: Changes in Quality of Life (as Measured With the PAVK 86 Questionnaire) From Baseline to the End of Period 3
Description: as for outcome 13
Time Frame: From Baseline to the end of 6-months Follow-up (Period 3)
Population: Full Analysis Set (FAS). For each subscale of the questionnaire, Mean and SD are presented for non-missing values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alprostadil | Pentoxifylline
Number analyzed (Participants) | 269 | 272
units on a scale
  Pain | -0.28 (0.57) | -0.41 (0.58)
  Functional status | -0.26 (0.58) | -0.35 (0.57)
  Anxiety | -0.20 (0.64) | -0.22 (0.66)
  Mood | -0.06 (0.48) | -0.12 (0.53)
  Social life | -0.09 (0.43) | -0.04 (0.45)
  Expectation of treatment | 0.07 (0.51) | 0.11 (0.49)
  State of general health during the last week | -0.43 (1.83) | -0.48 (1.98)
  Quality of life during the last week | -0.36 (2.09) | -0.39 (2.20)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected up to 8 months (246 days) from the 1-week Run-in Period over the 8-weeks Treatment Period (4 weeks Daily Treatment, 4 weeks Interval Treatment) to the end of the 6-months Follow-up Period.
Description: Adverse Events refer to the Safety Set (SS). SS includes all randomized subjects who received at least one dose of trial medication.
  Subjects did not receive any dose of trial medication in the Run-in Period, so Adverse Events shown here refer to Treatment and Follow-Up Period.
Arm/Group | Alprostadil | Pentoxifylline
Serious Adverse Events (participants affected / at risk) | 19/276 | 17/285
Other Adverse Events (participants affected / at risk) | 60/276 | 55/285
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alprostadil (N=276) | Pentoxifylline (N=285)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 3 (3) | 1 (1)
Angina Pectoris (Cardiac disorders) | 2 (2) | 0 (0)
Left Ventricular Failure (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac Failure (Cardiac disorders) | 1 (1) | 0 (0)
Ischaemic Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial Flutter (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Failure Acute (Cardiac disorders) | 0 (0) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia Paroxysmal (Cardiac disorders) | 0 (0) | 1 (1)
Vestibular Disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Oedema Peripheral (General disorders) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 1 (1)
Device Related Infection (Infections and infestations) | 1 (1) | 0 (0)
Postoperative Wound Infection (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 1 (1)
Tinea Pedis (Infections and infestations) | 0 (0) | 1 (1)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cardiac Enzymes Increased (Investigations) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bronchial Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostatic Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carotid Artery Stenosis (Nervous system disorders) | 3 (3) | 0 (0)
Intercostal Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Suicide Attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Renal Failure Chronic (Renal and urinary disorders) | 0 (0) | 1 (1)
Genital Haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 4 (4) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
Extremity Necrosis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral Ischaemia (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alprostadil (N=276) | Pentoxifylline (N=285)
Angina Pectoris (Cardiac disorders) | 0 (0) | 4 (4)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 4 (5)
Abdominal Pain Upper (Gastrointestinal disorders) | 2 (2) | 6 (6)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 9 (10)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3)
Oedema Peripheral (General disorders) | 4 (4) | 2 (2)
Influenza Like Illness (General disorders) | 3 (3) | 5 (6)
Infusion Site Irritation (General disorders) | 3 (3) | 0 (0)
Infusion Site Swelling (General disorders) | 3 (4) | 0 (0)
Infusion Site Erythema (General disorders) | 2 (2) | 0 (0)
Infusion Site Extravasation (General disorders) | 0 (0) | 2 (4)
Infusion Site Haematoma (General disorders) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 3 (3) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2) | 3 (3)
Tooth Infection (Infections and infestations) | 2 (2) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Blood Creatinine Increased (Investigations) | 2 (2) | 0 (0)
Blood Glucose Increased (Investigations) | 2 (2) | 0 (0)
Transaminases Increased (Investigations) | 2 (2) | 0 (0)
Blood Pressure Increased (Investigations) | 0 (0) | 2 (2)
Blood Triglycerides Increased (Investigations) | 0 (0) | 3 (3)
Diabetes Mellitus (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 3 (3) | 4 (4)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Sleep Disorder (Psychiatric disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2)
Night Sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 4 (4) | 4 (4)
Flushing (Vascular disorders) | 3 (3) | 0 (0)
Phlebitis (Vascular disorders) | 2 (2) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days